CLINICAL TRIAL: NCT05686954
Title: Nutritional Effects of Different Doses of Cottonseed Oil in Humans
Brief Title: Cottonseed Oil Dose Response
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Collaborators: Cotton Incorporated (Unknown)
Responsible Party: Principal Investigator, Jamie Cooper, PhD, Professor, Director of UGA Obesity Initiative, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PROJECT00006633
Record Dates: First submitted 2023-01-05; First posted 2023-01-17 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Dyslipidemias; Overweight and Obesity; Nutrition, Healthy
MeSH Terms: conditions — Dyslipidemias; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Four groups of 28-day parallel feeding trials with three groups receiving different amounts of cottonseed oil (low, mid, high) and one group serving as control receiving a mixture of oils that match the fatty acid profile of the average American diet.
Who Masked: Participant
Masking Description: Participants are blinded to which group they are in and what oil they are receiving.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CSO LOW (Experimental): Participants are given foods enriched with cottonseed oil and instructed on how to substitute study foods into their diet to maintain caloric balance.
  Interventions: Other: CSO LOW
- CSO MID (Experimental): Participants are given foods enriched with cottonseed oil and instructed on how to substitute study foods into their diet to maintain caloric balance.
  Interventions: Other: CSO MID
- CSO HIGH (Experimental): Participants are given foods enriched with cottonseed oil and instructed on how to substitute study foods into their diet to maintain caloric balance.
  Interventions: Other: CSO HIGH
- CONTROL (Active Comparator): Participants are given foods enriched with a mixture of oils and instructed on how to substitute study foods into their diet to maintain caloric balance.
  Interventions: Other: CONTROL

INTERVENTIONS:
Other: CSO LOW — Participants are provided a breakfast shake and a snack daily that delivers 10% of the participant's estimated energy needs as cottonseed oil for 28 days.
  Arms: CSO LOW
Other: CSO MID — Participants are provided a breakfast shake and a snack daily that delivers 20% of the participant's estimated energy needs as cottonseed oil for 28 days.
  Arms: CSO MID
Other: CSO HIGH — Participants are provided a breakfast shake and a snack daily that delivers 30% of the participant's estimated energy needs as cottonseed oil for 28 days.
  Arms: CSO HIGH
Other: CONTROL — Participants are provided a breakfast shake and a snack daily that delivers 10% of the participant's estimated energy needs as a mixture of oils that match the average American fat intake for 28 days.
  Arms: CONTROL

SUMMARY:
Adding cottonseed oil to the diet has been shown to improve cholesterol profiles and other markers of chronic disease risk in both healthy and at-risk adults. However, CSO has only been tested in the context of high-fat diets. The goal of this clinical trial is to learn about the health effects of lower amounts of cottonseed oil (CSO) added to the diet in adults at increased risk for cardiovascular disease.

The main questions it aims to answer are:

* How do different amounts of CSO in the diet affect fasting cholesterol profiles and markers of liver function?
* How do different amounts of CSO in the diet affect fasting and post-meal markers of lipid metabolism (i.e. triglycerides) and glycemic control (i.e. blood sugar and insulin)?
* How do different amounts of CSO in the diet affect fasting and post-meal markers of chronic disease risk factors such as oxidative stress, inflammation, coagulation potential, and appetite control?

Participants will be asked to:

* Consume provided breakfast shakes and snacks daily for 28-days.
* Attend three weekly short visits for fasting blood draws, body measurements, and collect the next week of study materials.
* Attend two longer (5.5 h) testing visits which include eating a standardized breakfast meal and having blood drawn periodically before and after breakfast.

Researchers will compare CSO LOW, CSO MID, CSO HIGH, and Control groups (receiving a mixture of oils) to see if lower doses of CSO in the diet impart the same health benefits as previously shown with high doses of CSO.

DETAILED DESCRIPTION:
Cardiovascular disease risk factors, including higher BMIs and poor cholesterol profiles, are on the rise and contribute to the United States' growing disease burden. Cottonseed oil (CSO) is found readily in our food supply. Our previous studies have demonstrated that incorporating CSO into the diet is sufficient to reduce fasting total cholesterol (TC) and low-density lipoprotein cholesterol (LDL-c), increase high-density lipoprotein cholesterol (HDL-c), and improve postprandial lipid and/or glycemic responses in both healthy and at-risk populations. However, in these human studies, diets provided 30-44% of total energy from CSO, which corresponded to high-fat (HF) diet intake (40-50% of energy). The impact of lower doses of CSO on human health has yet to be tested. Therefore, this study aims to investigate whether lower doses of CSO are equally effective as previously proven high doses for improving fasting and postprandial lipid metabolism and markers of chronic disease risk. If lower doses of CSO in the diet are found to improve these markers, these study findings could lead to improvements in health.

This prospective clinical study is a single-blinded, randomized control trial in adults at increased risk for cardiovascular disease (poor cholesterol profiles or overweight/obesity). There are four diet interventions: CSO LOW (10% energy from CSO), CSO MID (20% energy from CSO), CSO HIGH (30% energy from CSO), and CON (10% energy from control oil mix). The study protocol consists of a 28-day intervention where participants are provided breakfast shakes and snacks that contain different amounts of cooking oil depending on their random group assignment.

There are a total of 6 testing visits: screening (v0), pre-intervention (v1), 3 weekly short visits (v2, v3, v4), and post-intervention (v5).

At screening (v0), qualification is confirmed based on anthropometrics and fasting blood draw, which is analyzed for a cholesterol panel and blood glucose. Additionally, energy requirements are estimated at this visit for use in the diet intervention.

At v1, participants will have anthropometrics measured, including body composition, by BodPod. Next, a certified phlebotomist places an IV catheter and takes the fasting blood sample. Then the participant consumes a high-saturated-fat meal challenge which delivers 35% of their estimated energy needs (from v0). Then the participant has blood drawn 8 times using the IV catheter over the next 5 hours.

28-day dietary intervention: Before leaving v1, participants are sent home with their first week's supply of daily shakes and snacks corresponding to their randomly assigned group. The ingredients for the breakfast shakes and snacks are identical between groups, the only difference being the amount of the assigned oil incorporated into the foods. All foods are portioned based on individual energy needs as estimated at v0.

Participants return weekly (v2, v3, v4) to return study materials and collect food for the next week. At these weekly visits, participants also have a fasting blood draw, body measures and consume their first breakfast shake of the week in the lab.

At the end of the 28-day dietary intervention, participants return for v5, where all procedures from v1 are repeated.

The investigators hypothesize that CSO LOW, CSO MID, and CSO HIGH will improve the proposed overall health outcomes and markers of chronic disease risk without changing inflammatory markers compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* 25-75-year-old men and women at increased risk for cardiovascular disease. Increased risk for cardiovascular disease will be defined by either elevated cholesterol profiles -or- overweight/obesity.
* Elevated cholesterol profiles will be defined as:
* "Borderline High" and/or "at risk" in two or more of the following variables (total cholesterol: 180-239 mg/dL, LDL cholesterol 110-159 mg/dL, triglycerides 130-199 mg/dL) --or---
* "High" in total cholesterol (240 mg/dL and higher), LDL (160 mg/dL or higher), or triglycerides (between 200 - 350 mg/dl).

Overweight/obesity will be defined by body mass index (overweight 25-29.9 kg/m2 or obesity 30 kg/m2 or greater).

Exclusion Criteria:

* Probable familial hypercholesterolemia, defined by: total cholesterol greater than 290 mg/dL or LDL levels greater than 190 mg/dL plus a family history of myocardial infarction (MI) before 50 years of age in a 2nd-degree relative or below age 60 in a 1st-degree relative.
* women on hormone replacement therapy for less than 2 years
* women who are pregnant
* individuals who regularly exercise more than 3 h/w
* weight gain or loss of more than 5% of their body weight in the past 3 months
* plans to begin a weight loss/exercise regimen during the trial
* history of medical or surgical events that could affect digestion or swallowing
* gastrointestinal surgeries, conditions or disorders,
* any chronic diseases (including moderate to severe asthma, chronic lung disease, and kidney disease),
* metabolic diseases
* atherosclerosis
* previous MI or stroke
* cancer
* fasting blood glucose levels greater than 126 mg/dL
* blood pressure greater than 180/120 mmHg
* medication use affecting digestion and absorption, metabolism (e.g., thyroid meds), lipid-lowering medications, medications for diabetes, steroid/hormone therapies, or current antibiotic cycles
* medically prescribed or special diets
* Food allergies (specific to the foods in the study, including wheat, dairy, and cottonseed oil)
* fish oil supplements,
* excessive alcohol use (greater than 3 drinks/d for men; greater than 2 drinks/d for women)
* tobacco or nicotine use
* underweight BMI (<18.5 kg/m2)

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change in fasting serum lipoprotein and cholesterol concentrations | baseline, 4 weeks
  The concentration of fasting serum total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, apolipoprotein B (mg/dl)
Change in fasting serum lipoprotein particle numbers | baseline, 4 weeks
  Number of particles of low density lipoproteins (LDL), LDL small, HDL large, LDL medium, lipoprotein (a) (nmol/L)
Change in fasting and postprandial plasma triglyceride concentrations | baseline, 4 weeks
  The concentration of plasma triglycerides before and after the high saturated fat meal challenge at both pre- and post-intervention visits (mg/dL)
Change in fasting and postprandial plasma non-esterified fatty acid (NEFA) concentrations | baseline, 4 weeks
  The concentration of plasma NEFAs before and after the high saturated fat meal challenge at both pre- and post-intervention visits (mEq/L)
Change in fasting and postprandial plasma glucose concentrations | baseline, 4 weeks
  The concentration of plasma glucose before and after the high saturated fat meal challenge at both pre- and post-intervention visits (mg/dL)
Change in fasting and postprandial plasma insulin concentrations | baseline, 4 weeks
  The concentration of plasma insulin before and after the high saturated fat meal challenge at both pre- and post-intervention visits (uU/mL)
Change in fasting and postprandial plasma appetite control hormones concentrations | baseline, 4 weeks
  The concentration of plasma appetite control hormones before and after the high saturated fat meal challenge at both pre- and post-intervention visits. Appetite control hormones include Cholecystokinin (CCK), Peptide YY (PYY), Ghrelin (pg/mL)
Change in fasting and postprandial subjective feelings related to appetite | baseline, 4 weeks
  Visual analog scale ratings of feelings related to appetite before and after the high saturated fat meal challenge at both pre- and post-intervention visits. Subjective feelings of hunger, fullness, desire to eat, prospective consumption, and a composite appetite score are measured by visual analog scales (mm).
Change in fasting and postprandial plasma Malondialdehyde (MDA) | baseline, 4 weeks
  The concentration of MDA before and after the high saturated fat meal challenge at both pre- and post-intervention visits (nmol/mL).
Change in fasting and postprandial plasma total antioxidant capacity | baseline, 4 weeks
  Total antioxidant capacity before and after the high saturated fat meal challenge at both pre- and post-intervention visits (U/mL).
Change in fasting and postprandial plasma inflammatory cytokine concentrations | baseline, 4 weeks
  The concentration of interleukin-1 beta, C reactive protein, tumor-necrosis factor-alpha, and interleukin-6 before and after the high saturated fat meal challenge at both pre- and post-intervention visits (pg/mL).
Change in fasting and postprandial plasma markers of coagulation potential | baseline, 4 weeks
  The concentration of plasminogen activator inhibitor-1, and tissue factor before and after the high saturated fat meal challenge at both pre- and post-intervention visits (pg/mL).
Change in fasting and postprandial plasma angiopoietin-like (ANGPTL) proteins | baseline, 4 weeks
  The concentration of ANGPTL 3, ANGPTL 4, and ANGPTL 8 before and after the high saturated fat meal challenge at both pre- and post-intervention visits (ng/mL).
Change in fasting insulin resistance metrics | baseline, 4 weeks
  Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) and Homeostatic Model Assessment for β-cell function (HOMA-B) will be calculated from fasting insulin and glucose measures before and after the 28-day intervention.

SECONDARY OUTCOMES:
Change in fasting serum hepatic enzymes | Baseline, 4 weeks
  Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Alkaline phosphatase (ALP), Gamma-Glutamyl Transferase (GGT) (U/L)
Change in fasting serum hepatic proteins | Baseline, 4 weeks
  Total protein and albumin (g/dL)
Change in fasting serum bilirubin | Baseline, 4 weeks
  Total total bilirubin, direct bilirubin, and indirect bilirubin (mg/dL)
Change in additional fasting and postprandial plasma appetite control hormones concentrations | baseline, 4 weeks
  The concentration of additional plasma appetite control hormones before and after the high saturated fat meal challenge at both pre- and post-intervention visits. Additional appetite control hormones include Glucagon-like peptide-1 (GLP-1), Gastric inhibitory peptide (GIP), Pancreatic Polypeptide (PP) (pg/mL)
Change in fasting and postprandial plasma antioxidant parameters | baseline, 4 weeks
  Glutathione peroxidase activity, superoxide dismutase activity, glutathione-s-transferase activity before and after the high saturated fat meal challenge at both pre- and post-intervention visits (U/mL).
Change in additional fasting and postprandial plasma inflammatory cytokine concentrations | baseline, 4 weeks
  The concentration of monocyte chemoattractant protein-1, and interleukin-10 before and after the high saturated fat meal challenge at both pre- and post-intervention visits (pg/mL).
Change in additional fasting and postprandial plasma markers of coagulation potential | baseline, 4 weeks
  The concentration of Von Willebrand factor, tissue factor pathway inhibitor, fibrinogen and D-dimer before and after the high saturated fat meal challenge at both pre- and post-intervention visits (pg/mL).
Change in acute dietary intake | baseline, 4 weeks
  One-day food logs will be used to record all foods and beverages consumed on testing days

OTHER OUTCOMES:
Change in blood pressure | baseline, 4 weeks
  Systolic and diastolic blood pressure (mmHg)
Change in body weight | baseline, 4 weeks
  body weight (kg)
Change in body composition | baseline, 4 weeks
  BodPod will be used to measure body fat percentage (body fat %)
Change in diet composition | baseline, week 2, week 4
  3-day food logs will be used to record foods and beverages consumed before and during the 28-day intervention period
Change in fasting and postprandial fatty acid composition | baseline, 4 weeks
  Fatty acid composition of plasma before and after the high saturated fat meal challenge at pre- and post-intervention visits (% total triglycerides).
Change in fasting tocopherol concentrations | baseline, 4 weeks
  Plasma tocopherol concentrations (ug/ml)
Change in anthropometric circumferences | baseline, 4 weeks
  hip and waist circumferences (cm)
Change in resting metabolic rate | Screening
  Resting metabolic rate (RMR) will be measured for 30 minutes on the TrueOne 2400 (Parvo Medics, Sandy, UT)
Change in perceived stress | baseline, 4 weeks
  Perceived Stress Scale will be administered and scored to determine stress levels
Change in anxiety | baseline, 4 weeks
  The State Trait Anxiety Inventory will be administered and scored to determine anxiety levels.
Change in self reported physical activity levels | baseline, 2 weeks, 4 weeks
  The International Physical Activity Questionnaire will be used to collect self-reported average physical activity levels (met/min)
Change in body Mass Index (BMI) | baseline, 4 weeks
  BMI will be calculated based on height and weight measures (kg/m2)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie A Cooper, Ph.D., Principal Investigator — University of Georgia
Locations (1):
- University of Georgia, Athens, Georgia, United States

REFERENCES:
- [Derived] Hawkins CD, Prater MC, Ward CA, Paton CM, Cooper JA. Dose-Response Effects of Cottonseed Oil on Blood Lipid Responses in Adults at Risk of Cardiovascular Disease: A Randomized Controlled Trial. J Nutr. 2025 Nov 12:S0022-3166(25)00702-3. doi: 10.1016/j.tjnut.2025.11.006. Online ahead of print. PMID 41238122